CLINICAL TRIAL: NCT03481504
Title: Study Protocol of a Single Case Methodology Experiement Exploring the Effectiveness and Feasibility of an Exposure-centered ACT Intervention for Chronic Pain Patients: A Pilot Study
Brief Title: A New Approach in Chronic Pain; Acceptance & Commitment Therapy-Exposure & Perspective Taking (ACT-EPT)
Acronym: ACT-EPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NL63888.068.17
Record Dates: First submitted 2018-03-19; First posted 2018-03-29 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Single case methodology with a multple baseline design in a mixed methods approach in which a quantitative approach will be followed by a qualitative approach. The star of the experiemental intervention will be randomized
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The particpant is kept naieve about the fact that the moment of starting the intervention is randomized but coiuld not be blinded for the intervention. The outcome assessor and investigator are blinded for randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-ETP (Experimental): Cognitive behavioral treatment
  Interventions: Behavioral: Acceptance & Commitment Therapy-Exposure and Perspective Taking
- Usual care (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Acceptance & Commitment Therapy-Exposure and Perspective Taking — To increase patients' participation by improving their level of coping with chronic pain.
  Arms: ACT-ETP

SUMMARY:
Background: Chronic pain is a highly prevalent phenomenon with a large impact on the individual's wellbeing. Acceptance and Commitment Therapy (ACT) can be used to help patients relate to chronic pain in a way that helps improve their quality of life. This paper introduces an ACT protocol specific to chronic pain patients: ACT- Exposure and Perspective Taking (ACT-EPT). Aspects specific to this therapy are the focus on exposure as a means to elicit behavioural and emotional change regarding pain experience and it's format as a compact individual therapy.

Objectives: Investigators conduct a single case experimental study (ABA design) with a multiple baseline design, aimed at assessing the effectiveness of the experimental ACT-EPT protocol (phase B) compared to usual care (phase A) in individual chronic pain patients. Outcomes include the increase of participation in daily life and health related quality of life, measured with the Short Form-12 (SF-12). Quantitative results will be combined with qualitative results from interviews in a mixed methods design.

Participants: Five adults with chronic pain referred to a rehabilitation centre (≥18 years old).

Methods: Phases A and B together take 16 weeks for each participant, during which weekly quantitative measurements will be taken. The length of the first phase A will be randomised. The intervention (phase B) consists of weekly ACT-EPT sessions with a maximum of 3 sessions of approximately 90 minutes each. Individual interviews will take place after the last quantitative measurements. These focus on two topics: psychological processes of change and evaluating the intervention.

DETAILED DESCRIPTION:
Rationale: Chronic pain is a phenomenon with a large impact on the individual's wellbeing and is a problem with a large global burden of disease, with a prevalence of 19 to 20% in European adults and an annual cost of €200 billion in Europe. Apart from causing physical suffering, chronic pain can lead to depression, suicidal thoughts and disrupted social relationships and can cause impairments in everyday life tasks and activities. Despite the seriousness of chronic pain, not all chronic pain patients receive adequate treatment. One cognitive behavioral therapy treatment which is used in the Netherlands for chronic pain patients is the Acceptance and Commitment Therapy (ACT). However, the way in which this therapy is delivered in the Netherlands tends to take many sessions. It therefore seems attractive to investigate a short version of this protocol, which was developed in Sweden. This short version, ACT-EPT, is already being used in the Netherlands on a small scale but its effects have not yet been studied. The current paper proposes a pilot study with an innovative N-of-1 design to investigate this therapy's effectiveness.

Objective: Investigating the effectiveness of an experimental protocol of Acceptance and Commitment Therapy-Exposure & Perspective Taking (ACT-EPT) compared to usual care in individual chronic pain patients on the increase of their participation in daily life and health related quality of life, as measured with the SF-12 in a study with a single case experimental methodology.

Study design: The randomized n=1 study combines a quantitative and a consecutive qualitative part (mixed methods). Each participant receives the intervention and serves as his or her own control in an AB design. In phase A, all participants continue the care they already received which will be recorded as their care as usual. At a random moment, phase A will end and participants will start their intervention, thus entering phase B. This study randomizes participants on the duration of phase A, which means that the lengths of phases A and B differs among participants. The total study period (A+B) over which participants will receive weekly measurements is the same for all participants (16 weeks). Results will be presented on an individual basis according to the single case experimental methodology. In the last week of the total period, participants will be invited for an interview with a researcher focussing on their experience living with chronic pain and to evaluate the intervention. This interview will take place in the participants' own environment. Methodological details of all aspects of the design will be explained further in the protocol.

Study population: Chronic pain patients of 18 years or older referred the Rehabilitation Centre Winnock Zorg in Heerlen or Arnhem for treatment (n=5).

Intervention: The ACT-EPT treatment protocol is a type of acceptance-based cognitive behavioral therapy, aimed to increase patients' participation by improving their level of coping with chronic pain. The therapy takes between one and three sessions of about an hour and a half each.

Main study parameters/endpoints: The primary outcome measure of this study is the SF-12. Secondary outcome measures are the AAQ-II-P, PIPS, PSK, PDI, NPRS , IPA, FFMQ-SF and the ELS. The PSK will only be used for clinical purposes.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: No risks are associated with this study. The load for the participants consists of the weekly filling out of a limited amount of questionnaires and the participation in a one hour interview. The number of questionnaires that patients are asked to fill out differs per week, with a lowest load per week of 8 minutes and the highest load at baseline of 55 minutes. The total time taken to fill out all questionnaires over the 16 week period is 6 hours and 55 minutes, with an average of 26 minutes per week. Detailed information can be found in the questionnaires table in the protocol. The intervention takes between one and three sessions of about an hour and a half each, and is given in the rehabilitation centre.

ELIGIBILITY:
Inclusion Criteria:

* The patient is diagnosed as having chronic pain, is referred to Winnock Zorg rehabilitation center, location Heerlen or Arnhem, and is registered to receive treatment at Winnock Zorg rehabilitation center;
* The patient has pain of the musculoskeletal system
* The patient has pain for longer than 6 weeks
* The patient is medically stable
* The patient has functional limitations
* The medical history and examination of the patient do not indicate further somatic diagnostics and treatment
* The patient has unwanted psychosocial consequences from the pain, such as in activities of daily life, relationships, work and social role
* Social and psychological factors are complex and play an important role in maintaining the pain, as is assessed by a rehabilitation physician expert
* The patient shows to have insights in his/her functional limitations, as is assessed by a rehabilitation physician expert
* The patient has an active attitude in finding solutions for his/her problem, as is assessed by a rehabilitation physician expert
* The assessment of the patient by a rehabilitation physician expert indicates that the patient is open to receive a cognitive therapy for pain management;
* The patient is at least 18 years old;

Exclusion Criteria:

* The patient has a history of diagnosed psychotic illness or manic episode;
* The patient has a diagnosed systematic or malignant disease;
* The patient has had a form of Acceptance and Commitment Therapy in the past;
* The patient is using a type of CBT at the moment of the study;
* The patient has a reported substance abuse within 6 months before the trial;
* The patient has a serious medical condition which can be expected to interfere with participation in the study.
* The patient has an inadequate understanding of the written and spoken Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
SF-12 | Change between all weekly time-points SF-12 until 16 weeks after randomisation will be calculated
  The SF-12 measures overall quality of life and includes items that assess participation. The SF-12 is a frequently used measure and has shown to have good internal consistency, reliability, construct validity and responsiveness in patients with chronic (low) back pain (Luo et al., 2003). The measure is a subset of 12 items from the SF-36 including 6 items from the physical summary measure (PCS) and 6 items from the mental summary measure (MCS).

CONTACTS AND LOCATIONS:
Locations (1):
- Winnock Zorg, Heerlen, Netherlands

IPD SHARING:
Plan to Share IPD: No